CLINICAL TRIAL: NCT03686787
Title: The Efficacy of Oral Tranexamic Acid and a 1927 nm Diode Laser in Patients With Melasma. A Prospective Randomized Split Face Study
Brief Title: Oral Tranexamic Acid and Laser for Treatment of Melasma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laser and Skin Surgery Center of New York (Other)
Collaborators: Dermatology & Laser Surgery Center, Houston, TX (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSSC-TA-CB-ASDS
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Melasma
Keywords: melasma; chloasma; tranexamic acid; nonablative laser resurfacing; sunscreen; hyperpigmentation
MeSH Terms: conditions — Melanosis; Hyperpigmentation | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Healthy, non-smoking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tranexamic Acid — A split face study of oral tranexamic acid in combination with laser treatment
  Other Names: 1927 nm nonablative laser

SUMMARY:
Tranexamic acid and 1927 diode laser non-ablative fractionated laser for the treatment of Melasma.

DETAILED DESCRIPTION:
Seeking healthy non-smoking male and female volunteers of all skin types of age 18 to 50 with moderate melasma or severe melasma. Participants will receive up to 5 monthly laser treatments to half the face and need to take a pill twice a day for 4 months. Follow up visits are required 1 month, 3 months and 6 months after the final treatment. Compensation of up to $150 will be provided based on completed visits.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 50 Skin types I through VI (all skin types) Moderate or severe melasma

Exclusion Criteria:

Pregnant or nursing women Current use of hormonal birth control medication or any hormonal therapy Use of topical steroids within 1 month of study enrollment Use of topical hydroquinone within 3 months of study enrollment History of laser or dermabrasion to the face within 6 months of study enrollment Regular use of tanning parlors Occupation involving primarily outdoor activities Current treatment with blood thinning medications History of thrombosis or thrombophilia History of thromboembolic disease, such as deep vein thrombosis, pulmonary embolism and/or cerebral thrombosis Family history of thromboembolic disease History of stroke History of >2 spontaneous abortions History of kidney dysfunction History of cancer Smoking Significant cardiovascular or respiratory disease (end-stage congestive heart failure or chronic obstructive pulmonary disease) History of subarachnoid hemorrhage History of acquired disturbances of color vision Known allergy to tranexamic acid As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of mMASI (Modified Melasma Area and Severity Index) | 16 weeks
  The difference between mMASI at week 0 and mMASI at week 16

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Laser & Skin Surgery Center of New York, New York, New York
  - Dermatology & Laser Surgery Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.laserskinsurgery.com